CLINICAL TRIAL: NCT06075212
Title: Immune Reconstitution After Allogeneic Hematopoietic Stem Cell Transplantation With Post-transplant Blinatumomab Maintenance Treatment
Brief Title: Immune Reconstitution After Allo-HSCT and Blinatumomab
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Principle Investigator, Sichuan University
Other Study IDs: Blin-immune 1.0
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Leukemia, Lymphoid
MeSH Terms: conditions — Leukemia, Lymphoid | interventions — blinatumomab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Blin-PTCY: Post-transplant cyclophosphamide is used as graft versus host disease (GvHD) prophylaxis. Treatment with blinatumomab was initiated within 60 to 90 days after transplantation and was administered bimonthly until 1 year after transplantation.
  Interventions: Drug: blinatumomab
- Blin-ATG: Antithymocyte globulin is used as graft versus host disease (GvHD) prophylaxis. Treatment with blinatumomab was initiated within 60 to 90 days after transplantation and was administered bimonthly until 1 year after transplantation.
  Interventions: Drug: blinatumomab
- Control: Patients don't take blinatumomab treatment after transplantation.

INTERVENTIONS:
Drug: blinatumomab — The dose of one course was as follows: day 1-2: 8ug/day, continuous intravenous drip for 24 hours, day 3-7: 16ug/day, continuous intravenous drip for 24 hours. Treatment with blinatumomab was initiated within 60 to 90 days after transplantation and was administered bimonthly until 1 year after transplantation. Dexamethasone 20mg was administered 1 hour before administration on days 1 and 3 to prevent adverse events.
  Groups: Blin-ATG; Blin-PTCY

SUMMARY:
The goal of this observation study is to test in relapsed or refractory acute lymphoblastic leukemia (R/R ALL) patients undergoing allogeneic hemopoietic stem-cell transplantation (allo-HSCT). The main question it aims to answer is:

• Effect of post-transplant blinatumomab treatment on immune reconstitution after transplantation.

Participants will undergo immune repertoire sequencing(IR-SEQ) before blinatumomab treatment, 6 months and 1 year after transplantation.

Researchers will compare patients who don't receive blinatumomab treatment after transplantation to see if TCR or BCR expression differs.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16-65 years old
2. KPS score > 60 or ECOG score 0-2
3. diagnosed as B-ALL, a) disease status > CR1 at the time of transplantation; Patients beyond CR1 or induction failure could be free of minimal residual disease (MRD). b) any residual disease, defined as >0.01% leukemic cells by flow cytometry, BCR-ABL transcript ≥ 1 in 10000 by PCR, or high-risk genetic abnormality
4. neutrophil count ≥0.5×10^9/L and platelet count ≥20×10^9/L
5. creatinine clearance ≥30ml/min; Alanine aminotransferase/aspartate aminotransferase ≤5 times the upper detection limit; Total bilirubin ≤3 times the upper limit of detection
6. The first initiation of berintuzumab therapy was within 60-100 days after transplantation
7. without evidence of active acute graft-versus-host disease (aGvHD)

Exclusion Criteria:

1. With serious basic diseases of important organs, such as myocardial infarction, chronic cardiac insufficiency, decompensated liver dysfunction, renal dysfunction, gastrointestinal dysfunction, etc
2. With clinically uncontrolled active infection
3. Patients with central nervous system involvement before transplantation
4. Poor graft function (PGF) occurred after allo-HSCT
5. Patients with second allogeneic transplantation

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Relapsed or refractory acute lymphoblastic leukemia (R/R ALL) patients undergoing allogeneic hemopoietic stem-cell transplantation (allo-HSCT).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
T cell receptor expression | before blinatumomab treatment , 6 months and 1 year
  T cell receptor expression measured by Immune Repertoire sequencing(IR-SEQ)
B cell receptor expression | before blinatumomab treatment , 6 months and 1 year
  B cell receptor expression measured by Immune Repertoire sequencing(IR-SEQ)

SECONDARY OUTCOMES:
T cell subsets count | before blinatumomab treatment , 6 months and 1 year
  T cell subsets count including CD3+, CD4+, CD8+, CD19+, Treg, memory and cytotoxic T cells

IPD SHARING:
Plan to Share IPD: No